CLINICAL TRIAL: NCT06364722
Title: Effect of Acupuncture on the Microbiota-gut-brain Axis in Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2024-02
Record Dates: First submitted 2024-03-29; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease
Keywords: acupuncture; brain-gut interaction
MeSH Terms: conditions — Crohn Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects, efficacy assessors and statisticians were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Subjects in this group will receive real acupuncture combined with real moxibustion.
  Interventions: Other: Acupuncture treatment
- Sham group (Sham Comparator): Subjects in this group will receive sham acupuncture combined with sham moxibustion.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture treatment — We selected acupoints including Zhongwan (CV12) and bilateral Shangjuxu (ST37), Sanyinjiao (SP6), Gongsun (SP4), Taichong (LR3), Taixi (KI3), Hegu (LI4), and Quchi (LI11)17 according to the World Health Organization standard. Single-use 0.30×40 mm or 0.30×25 mm acupuncture needles (Hwato, Suzhou, China) 27,28 were vertically inserted into each acupoint to 20-30 mm depth to obtain a deqi sensation (a soreness, distention, numbness or heaviness sensation). Bilateral Zusanli (ST36) and Tianshu (ST25) were selected for moxibustion. Pure moxa sticks (diameter: 2.8 cm; Hanyi, Nanyang, China) were ignited and fixed on a moxibustion stand at a distance of 3-5 cm to the surface of acupoints. The temperature of skin surface at the acupoints was maintained at 43 ± 1°C and monitored with a miniature infrared thermometer (Fluke 62, Fluke Corporation, Everett, WA, USA). Acupuncture and moxibustion were concomitantly performed for 30 min.
  Arms: Acupuncture group
Other: Sham acupuncture — Sham acupuncture needles (0.35×40 mm) with flat tips (Hwato, Suzhou, China) were inserted towards the same acupoints to induce slight pain but without penetrating the skin. Sham moxibustion was made by igniting the same type of moxa sticks but fixing them at a distance of 8-10 cm from the skin of acupoints to maintain the temperature at 37 ± 1°C. Sham acupuncture and moxibustion were concomitantly performed for 30 min.
  Arms: Sham group

SUMMARY:
Multidisciplinary techniques such as multimodal neuroimaging, microbiology, and bioinformatics were applied to study the differences in correlation characteristics between gut microbes, functional brain networks, and peripheral inflammation among patients with active Crohn's disease (CD), CD in remission, and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ age ≤ 75 years, gender is not limited;
2. Disease in mildly or moderately active stage: 150 ≤ CDAI < 450 and at least one of the following is met: serum C-reactive protein ≥ 5 mg/L, faecal calreticulin ≥ 250 μg/g, or endoscopic ulceration, or remission stage: CDAI < 150 and at least one of the following is met: serum C-reactive protein < 5 mg/L, faecal calreticulin < 250 μg/g, or endoscopic No ulcers;
3. Not taking or taking the following medications: mesalazine (≤4 g/d and have been taking for ≥1 month), prednisone (≤15 mg/d and have been taking for ≥1 month), and/or azathioprine (≤1 mg/kg/d and have been taking for ≥3 months);
4. Those who have not used biologics within 3 months prior to study entry;
5. Those who have never received acupuncture treatment;
6. Understand, agree to participate in the study and sign an informed consent form.

Exclusion Criteria:

1. Patients who have recently prepared for pregnancy or are pregnant or breastfeeding;
2. Patients with severe organic pathology;
3. Patients with confirmed psychosis;
4. Patients who are suffering from multiple diseases at the same time and taking other drugs for a long time which may affect the observation of this clinical trial;
5. Patients with severe extra-intestinal manifestations such as severe skin diseases (e.g., erythema nodosum, gangrenous pyoderma, etc.), ocular lesions (e.g., iritis, uveitis, etc.), and thromboembolic diseases;
6. Those with severe intestinal fistulae, abdominal abscesses, intestinal stenosis and intestinal obstruction, perianal lesions (perianal abscesses, etc.), gastrointestinal haemorrhage, intestinal perforation and other complications;
7. Those suffering from short bowel syndrome, those who have undergone abdominal or gastrointestinal surgery within the last six months;
8. Those who are unable to perform acupuncture due to the presence of skin diseases or defects in the area selected for acupuncture.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Effect of Acupuncture on Crohn's Disease Activity Index (CDAI) | Week 12
  Difference in Crohn's Disease Activity Index (CDAI) from baseline at 12 weeks was used for between-group assessment.

SECONDARY OUTCOMES:
Effects of Acupuncture on Anxiety and Depression | Week 12
  Differences in Hospital Anxiety Depression Scale (HADS) scores from baseline at 12 weeks were used for between-group assessment.
Effects of Acupuncture on Quality of Life | Week 12
  Differences in Inflammatory Bowel Disease Questionnaire (IBDQ) scores from baseline at 12 weeks were used for between-group assessment.
Effect of acupuncture on intestinal inflammation | Week 12
  Differences in serum C-reactive protein levels and faecal calprotectin levels from baseline at 12 weeks were used for between-group assessment.
Effects of acupuncture on gut microbiota | Week 12
  This includes the alpha and beta diversity of gut microbes and the abundance of flora at each level.
Effects of acupuncture on the functional activity of brain networks | Week 12
  Including brain network graph theory properties, connection strength.
Effects of acupuncture on intestinal inflammation | Week 12
  Including intestinal barrier function, peripheral Th1/Th17-related inflammatory factors.
Effect of Acupuncture on Brain Imaging-Gut Microbiological Correlations | Week 12
  The effect of acupuncture was observed by constructing correlations between brain imaging parameters and gut microbiology and gut inflammation levels.
Safety evaluation (number of participants with abnormal reactions to acupuncture and moxibustion treatment) | Week 12
  Abnormal reactions after acupuncture and moxibustion, such as bleeding, hematoma, scald, dizziness and other phenomena.
Safety evaluation (number of participants with abnormal routine blood tests) | Week 12
  Routine blood tests, which mainly include the number of red blood cells, white blood cells and platelets per litre of blood.
Safety evaluation (number of participants with abnormal Liver function tests) | Week 12
  Liver function tests, mainly including peripheral blood concentrations of alanine aminotransferase (U/L), glutamine aminotransferase (U/L), gamma-glutamyl transpeptidase (U/L), alkaline phosphatase (U/L), total bilirubin (μmol/L), direct bilirubin (μmol/L), indirect bilirubin (μmol/L), total protein (g/L), albumin (g/L) and globulin (g/L).
Safety evaluation (number of participants with abnormal Renal function tests) | Week 12
  Renal function tests, mainly including tests of creatinine (μmol/L) and urea nitrogen (mmol/L) concentrations in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, PhD, MD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian

IPD SHARING:
Plan to Share IPD: No